CLINICAL TRIAL: NCT06702800
Title: Clinical Exploratory Study on Predicting Drug Sensitivity for Breast Cancer Treatment Using Simulated Organoid Models.
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 1106852441
Record Dates: First submitted 2024-09-14; First posted 2024-11-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Consist of tumor tissue samples obtained by puncture from patients with advanced breast cancer and 5 ml of venous blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this trial, we plan to construct a patient-derived organoid (PDO) model using fresh tumor tissue samples. Taking the relevant data of drug efficacy of breast cancer organoids as an example, it is shown that organoids may provide predictive information for drug sensitivity and may improve the therapeutic effect of advanced tumors. In this way, we aim to verify the effectiveness, feasibility and consistency of the PDO model in predicting treatment, and establish an evaluation system for treatment plans to help precision treatment of breast cancer.

DETAILED DESCRIPTION:
This study is a prospective, observational clinical research focusing on the drug sensitivity of patient-derived organoid (PDO) models, aiming to evaluate the consistency between the drug sensitivity of PDO models and the efficacy of selected clinical regimens.

1. Primary endpoint: The consistency between the drug sensitivity of the PDO model in analyzing treatment regimens and the objective response rate (ORR) of patients in clinical treatment.
2. Secondary endpoints: 1. To determine whether the PDO model can highly replicate the characteristics of the tumor microenvironment and maintain a high degree of consistency with tumor tissues in terms of molecules, cells, and tissue structures.

2. Based on the collection of drug sensitivity results of PDO and clinical treatment data, to comprehensively analyze the statistical differences in progression-free survival (PFS), overall survival (OS), and disease control rates (DCR) between patients whose clinical treatment regimens are consistent with the drug sensitivity results of PDO and those who are not.

(3) Exploratory endpoints: 1. To conduct peripheral blood mononuclear cell (PBMC) isolation tests and RNA sequencing (RNA seq) for the included subjects, analyze the potential reasons for the differences in the consistency of PDO's predicted efficacy, and explore the underlying mechanisms.

2. To evaluate the effectiveness of the organoid model in predicting the drug sensitivity of subsequent treatments for early refractory breast cancer patients, that is, to analyze the consistency between the drug sensitivity results detected by the organoid model and the pathological complete response rate (pCR) of patients who actually received subsequent treatments.

3. To assess the accuracy of the organoid model in predicting the drug sensitivity results of HER-2 positive breast cancer patients and their consistency with subsequent treatments.

4. To detect the expression of Trop-2 in triple-negative breast cancer (TNBC) organoids and the drug sensitivity test results of gossatumab, Dato-DXd, and SKB264 through immunohistochemistry and other techniques, and to determine whether they are consistent with the clinical treatment efficacy; whether the low expression of Trop-2 in breast cancer organoids is related to drug resistance in the source patients.

(III) Research Contents:

1. Screen breast cancer patients who meet the inclusion and exclusion criteria, perform puncture sampling for organoid model culture and preparation, and identify and verify whether the breast cancer organoids match the histological type of the original tumor.
2. Evaluate drug sensitivity using organoid model culture technology.
3. Conduct tumor assessment every 6 cycles, regularly perform safety visits and record, and explore the consistency between the drug sensitivity evaluated by the organoid model culture technology and the actual therapeutic effect of clinical patients, as well as the effectiveness and safety of this protocol.

3.1 Establishment of a PDO culture system suitable for breast cancer This study will use the hanging drop method organoid culture system, which can better preserve the tumor microenvironment of tumor cells, for the experiment. Breast cancer puncture samples obtained through informed consent will be digested into single-cell suspensions for organoid culture. Successfully cultured organoids will be collected for PBMC and RNA seq detection to assess the consistency of organoid tissue characteristics with those of the patient's pathological tissue and the infiltration of immune cells and drug penetration in the hanging drop method organoids. In this way, we will establish that the hanging drop method organoids reproduce the histological characteristics and marker expression of the original tumor tissue.

3.2 Detection of patient sensitivity to different induction chemotherapy regimens using the PDO system Based on the PDO organoid culture system established above, we will culture organoids from samples that meet the inclusion criteria. Once the culture is successful, the organoids will be immediately treated with multiple chemotherapy regimens and the treatment regimens that the patients will receive. The cell viability of the organoids will be measured as an indicator of organoid survival. By directly comparing with the CellTiter-Glo3D cell viability assay, the sensitivity of the organoids to different chemotherapy regimens will be statistically analyzed, and the most sensitive treatment regimen will be screened out.

3.3 Collection of clinical data and consistency analysis of drug sensitivity test results This trial aims to complete drug sensitivity tests on 30 samples. According to the actual clinical treatment regimens, the data of the 30 samples will be divided into two groups: consistent or inconsistent with the best drug sensitivity test regimen. The differences in objective response rate and disease control rate between the two groups will be statistically analyzed. At the same time, based on the drug sensitivity screening results, the consistency of clinical efficacy indicators of these patients will be statistically analyzed. In terms of prognosis, the differences in overall survival and progression-free survival between the two groups will be statistically analyzed.

ELIGIBILITY:
1. Inclusion and Exclusion Criteria for Early - stage Breast Cancer 1.1 Inclusion Criteria Age between 18 and 70 years old, regardless of gender. ECOG score: 0 - 1. Clinically diagnosed or pathologically confirmed as breast cancer. TNM stage is T2 - 3 and Nx, and is currently receiving or planning to receive subsequent neoadjuvant therapy (including but not limited to chemotherapy, targeted therapy, endocrine therapy, etc.).

   According to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), there is at least one measurable lesion; the expected survival time is ≥ 12 weeks.

   The subject must recover from all toxicities caused by previous treatments (recovery to ≤ grade 1, evaluated based on CTCAE 5.0, or meet the inclusion criteria of the protocol), except for alopecia, vitiligo, or hypothyroidism that remains stable after hormone replacement therapy. (Note: For subjects with some chronic and stable grade 2 toxicities that the researcher deems related to previous anti - tumor treatments (such as chemotherapy - induced neuropathy), a decision on whether to include the subject in this study will be made after discussion with the medical monitor.) For female subjects with child - bearing potential and male subjects whose partners have reproductive potential, effective medical contraceptive measures should be taken during the research treatment period and within 6 months after the end of drug administration.

   Voluntarily sign the informed consent form, and be willing and able to comply with the follow - up, treatment, laboratory tests, and other research requirements specified in the research schedule.

   1.2 Exclusion Criteria Central nervous system (CNS) metastasis or carcinomatous meningitis. Bilateral breast cancer. History of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS). History of invasive breast cancer or metastatic breast cancer. Arterial or venous thrombosis events, such as deep vein thrombosis and pulmonary embolism, occurred within 3 months before randomization.

   Positive human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.

   Other serious diseases that are judged to potentially affect follow - up and short - term survival of the patient.

   Inability to swallow, chronic diarrhea, and intestinal obstruction, with various factors affecting drug intake and absorption.

   Known allergy to the potentially used treatment drugs. Adverse reactions of grade ≥ 1 that are still ongoing due to previous treatments. Exceptions are alopecia or cases that the researcher deems should not be excluded. Such cases should be clearly recorded in the investigator's notes.

   Female patients who are pregnant, breastfeeding, or planning to become pregnant during the study period (pregnancy tests should be considered for sexually active women of child - bearing age).

   Having had other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.

   Urinalysis shows urine protein ≥ 2+ or confirmed 24 - hour urine protein quantification > 1.0g; presence of any autoimmune diseases that still require treatment or a history of autoimmune diseases, excluding hypothyroidism caused by autoimmune thyroiditis that only requires hormone replacement therapy and type 1 diabetes with controllable and stable blood sugar.

   Patients with hypertension that cannot be well - controlled with a single antihypertensive drug (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); history of unstable angina pectoris; newly diagnosed angina pectoris within 3 months before screening or myocardial infarction event within 6 months before screening; arrhythmia (including QTcF: ≥ 450 ms for men and ≥ 470 ms for women) requiring long - term use of anti - arrhythmic drugs and New York Heart Association class ≥ II heart failure.

   Other situations that researchers evaluate as potentially endangering the patient's safety or having poor compliance, such as having serious diseases (including mental diseases), severely abnormal test results, and other high - risk factors in the family or society.
2. Inclusion and Exclusion Criteria for Advanced - stage Breast Cancer 2.1 Inclusion Criteria Age between 18 and 70 years old, both men and women are eligible. ECOG score: 0 - 1. Clinically or pathologically clearly diagnosed as advanced - stage breast cancer, regardless of molecular subtype.

   Currently receiving or planning to receive anti - tumor drug treatment, regardless of the number of treatment lines.

   According to the Response Evaluation Criteria in Solid Tumors (RECIST1.1), there is at least one measurable lesion; the expected survival time is ≥ 12 weeks.

   The subject must recover from all toxicities caused by previous treatments (recovery to ≤ grade 1, evaluated based on CTCAE5.0, or meet the inclusion criteria of the protocol), except for alopecia, vitiligo, or hypothyroidism that remains stable after hormone replacement therapy.

   (Note: For subjects with some chronic and stable grade 2 toxicities that the researcher deems related to previous anti - tumor treatments (such as chemotherapy - induced neuropathy), a decision on whether to include the subject in this study will be made after discussion with the medical monitor.) For female subjects with child - bearing potential and male subjects whose partners have reproductive potential, effective medical contraceptive measures should be taken during the research treatment period and within 6 months after the end of drug administration.

   Voluntarily sign the informed consent form, and be willing and able to comply with the follow - up, treatment, laboratory tests, and other research requirements specified in the research schedule.

   2.2 Exclusion Criteria Central nervous system (CNS) metastasis or carcinomatous meningitis. History of gastrointestinal perforation or fistula within half a year before medication or having a high bleeding risk.

   Positive human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.

   Other serious diseases that are judged to potentially affect follow - up and may lead to short - term survival of the patient.

   Inability to swallow, chronic diarrhea, and intestinal obstruction, with various factors affecting drug intake and absorption.

   Known allergy to the potentially used treatment drugs. Adverse reactions of grade ≥ 1 that are still ongoing due to previous treatments. Exceptions are alopecia or cases that the researcher deems should not be excluded. Such cases should be clearly recorded in the investigator's notes.

   Pregnant or breastfeeding women (pregnancy tests should be considered for sexually active women of child - bearing age).

   Having had other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.

   Occurrence of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 28 days before participating in this study.

   Urinalysis shows urine protein ≥ ++ or confirmed 24 - hour urine protein quantification > 1.0g.

   Patients with hypertension that cannot be reduced to the normal range with antihypertensive drugs (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg).

   Other situations that researchers evaluate as potentially endangering the patient's safety or having poor compliance, such as having serious diseases (including mental diseases), severely abnormal test results, and other high - risk factors in the family or society.
3. Criteria for Sample Exclusion

If a test sample meets any of the following criteria, it must be excluded:

Samples with unsuccessful PDO culture. Samples contaminated or failed due to improper operation during the test. Samples with lost data. Samples from patients who withdraw their informed consent and do not want to leave their samples.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR). | 2024-06-02 to 2026-05-31
  The proportion defined as subjects with complete remission (CR) and partial remission (PR) among all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No